CLINICAL TRIAL: NCT02535338
Title: A Phase 1/2 Trial of Erlotinib and Onalespib Lactate in EGFR-Mutant Non-Small Cell Lung Cancer
Brief Title: Erlotinib Hydrochloride and Onalespib Lactate in Treating Patients With Recurrent or Metastatic EGFR-Mutant Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01411; NCI-2015-01411 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-80; 9878 (Other: City of Hope Comprehensive Cancer Center LAO); 9878 (Other: CTEP); N01CM00038 (NIH); UM1CA186717 (NIH)
Record Dates: First submitted 2015-08-27; First posted 2015-08-28 (Estimated); Results first posted 2022-06-22 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (erlotinib hydrochloride, onalespib lactate) (Experimental): Patients receive erlotinib hydrochloride PO daily and onalespib lactate IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Onalespib Lactate; Other: Pharmacological Study

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: CP 358; CP-358; Cp-358,774; CP358; OSI 774; OSI-774; OSI774; Tarceva
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Onalespib Lactate — Given IV
  Other Names: AT-13387 Lactate; ATI-13387A; ATI-13387AU
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of onalespib lactate when given together with erlotinib hydrochloride and to see how well they work in treating patients with EGFR-mutant non-small cell lung cancer that has come back (recurrent) or has spread to other places in the body (metastatic). Erlotinib hydrochloride and onalespib lactate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of erlotinib hydrochloride (erlotinib) and onalespib lactate (onalespib) in patients with EGFR-mutant non-small cell lung cancer (NSCLC). (PHASE I) II. To preliminarily assess efficacy of combination erlotinib and onalespib at the recommended phase II dose (RP2D) determined in the phase I portion of the study in EGFR-mutant NSCLC patients who have not had a complete or partial response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 to frontline erlotinib after a minimum of 12 weeks on erlotinib. (PHASE II, COHORT A) III. To preliminarily assess efficacy of combination erlotinib and onalespib at the RP2D in NSCLC patients whose tumor harbors an EGFR exon 20 insertion (an EGFR mutation not typically responsive to single agent erlotinib). (PHASE II, COHORT B)

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity (primary aim phase II, secondary aim phase I).

II. To evaluate in a preliminary manner the progression-free survival (PFS) and disease control rate (DCR) of patients treated with erlotinib/onalespib.

III. To characterize the pharmacokinetics of the above drug combinations at the recommended phase II dose (RP2D).

TERTIARY OBJECTIVES:

I. To explore plasma EGFR-mutant deoxyribonucleic acid (DNA) as a biomarker by detecting changes in plasma EGFR-mutant DNA levels (including plasma EGFR-T790M) and new mutations that may represent resistance to treatment.

II. To demonstrate knockdown of Hsp90 client oncoproteins via treatment with erlotinib and onalespib by multiplexed immunofluorescence in serial tumor biopsies.

III. To establish patient derived xenotransplant models in EGFR-mutated NSCLC with a focus on tumors that lack response to single agent erlotinib and in patients with tumors harboring EGFR exon 20 insertions.

OUTLINE: This is a phase I, dose-escalation study of onalespib lactate followed by a phase II study.

Patients receive erlotinib hydrochloride orally (PO) daily and onalespib lactate intravenously (IV) over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for 1 year and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I: Patients must have metastatic/recurrent, histologically confirmed NSCLC that harbors an EGFR activating mutation (exon 21 L858R, exon 19 deletion, exon 18 G719X, exon 21 L861Q) with progressive disease by RECIST 1.1 on a previous EGFR-tyrosine kinase inhibitor (TKI); OR patients must have metastatic/recurrent histologically confirmed NSCLC that harbors an EGFR exon 20 insertion with progressive disease on platinum containing chemotherapy
* PHASE II COHORT A: Patients must have metastatic/recurrent histologically confirmed NSCLC that harbors an EGFR activating mutation (exon 21 L858R, exon 19 deletion, exon 18 G719X, exon 21 L861Q) with stable disease by RECIST 1.1 as best response on erlotinib compared to pre-treatment erlotinib imaging by RECIST 1.1 or progressive disease compared to pre-treatment imaging by RECIST 1.1 after a minimum duration of treatment on erlotinib of 12-weeks; patients must be enrolled within 6 months of initiation of erlotinib
* PHASE II COHORT B: Patients must have metastatic/recurrent histologically confirmed NSCLC that harbors an EGFR exon 20 insertion with progressive disease on or after platinum doublet chemotherapy
* FOR PHASE I: If patient is on erlotinib at the time of signed consent, the patient does NOT need to be discontinued prior to initiation of erlotinib and onalespib; other EGFR-TKIs must be discontinued at least 7 days prior to initiation of erlotinib and onalespib
* FOR PHASE II COHORT A: If patient is on erlotinib at the time of signed consent, erlotinib does NOT need to be discontinued prior to receiving treatment erlotinib and onalespib; last dose of erlotinib must be less than 28 days from when patient signs consent
* FOR PHASE II COHORT B: (EGFR exon 20 insertions): Prior EGFR-TKIs including erlotinib is allowed; if patient is on erlotinib at the time of signed consent, erlotinib does NOT need to be discontinued prior to initiation of erlotinib and onalespib
* Local testing for EGFR-mutations for this study is acceptable provided it was performed in a Clinical Laboratory Improvement Act (CLIA) certified lab
* Patients with a prior history of brain metastases are eligible provided:

  * The brain metastases have been treated
  * The patient is asymptomatic from the brain metastases
  * Corticosteroids prescribed for the management of brain metastases have been discontinued at least 7 days prior to registration
* Patients must have completed last chemotherapy >= 3 weeks or radiotherapy >= 2 weeks prior to receiving study drugs
* Patients must have recovered from adverse events attributable to previous treatment to =< grade 1, except for alopecia and sensory neuropathy =< grade 2
* Measurable disease by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) < 1.3 upper limit of normal (ULN)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of erlotinib and/or onalespib administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib and/or onalespib
* History of pneumonitis attributed to an EGFR inhibitor; history of radiation pneumonitis is allowed provided steroid administration for pneumonitis was not required
* Mean resting corrected QT interval (QTc using Fridericia's formula [QTcF]) > 470 msec
* Left ventricular ejection fraction =< 50% as demonstrated by echocardiogram or multigated acquisition scan (MUGA)
* Drugs that are known to increase torsades de pointes should be avoided; patients must discontinue these medications prior to enrollment on study; selection of alternate concomitant medications with no or minimal torsades de pointes potential is recommended
* Strong CYP3A4 inducers and inhibitors should be avoided; selection of alternate concomitant medications with no or minimal CYP3A4 enzyme inhibition potential is recommended; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with erlotinib and onalespib
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Prior treatment with a Hsp90 inhibitor
* Treatment with proton pump inhibitors within 3 days prior to study entry; if treatment with an histamine (H2)-receptor antagonist such as ranitidine is required, erlotinib must be taken 10 hours after the H2-receptor antagonist dosing and at least 2 hours before the next dose of the H2-receptor antagonist; although the effect of antacids on erlotinib pharmacokinetics has not been evaluated, the antacid dose and the erlotinib dose should be separated by several hours, if an antacid is necessary
* Abnormalities of the cornea based on history (e.g., dry eye syndrome, Sjogren's syndrome), congenital abnormality (e.g., Fuch's dystrophy), abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal Rose), and/or an abnormal corneal sensitivity test (Schirmer test or similar tear production test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Riess, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (6):
- United States (6):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California

REFERENCES:
- [Derived] Riess JW, Reckamp KL, Frankel P, Longmate J, Kelly KA, Gandara DR, Weipert CM, Raymond VM, Keer HN, Mack PC, Newman EM, Lara PN Jr. Erlotinib and Onalespib Lactate Focused on EGFR Exon 20 Insertion Non-Small Cell Lung Cancer (NSCLC): A California Cancer Consortium Phase I/II Trial (NCI 9878). Clin Lung Cancer. 2021 Nov;22(6):541-548. doi: 10.1016/j.cllc.2021.05.001. Epub 2021 May 15. PMID 34140248

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 - Onalespib IV 150 mg/m2; Dose Level -1 - Onalespib IV 120 mg/m2: Patients receive 150 mg erlotinib hydrochloride PO daily and onalespib lactate IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.
  Erlotinib Hydrochloride: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Onalespib Lactate: Given IV
  Pharmacological Study: Correlative studies
Period: Overall Study
Arm/Group | Dose Level 1 - Onalespib IV 150 mg/m2 | Dose Level -1 - Onalespib IV 120 mg/m2
Started | 3 | 8
Completed | 3 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 - Onalespib IV 150 mg/m2 | Dose Level -1 - Onalespib IV 120 mg/m2 | Total
Number analyzed (Participants) | 3 | 8 | 11
Age, Continuous [Median (Full Range); unit: years] | 51 [51 to 68] | 62.5 [53 to 70] | 60 [51 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1 | 6 | 7
  Asian | 1 | 1 | 2
  Hispanic | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 8 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Dose Limiting Toxicity (DLT)
Description: Adverse events were graded by CTCAE, v4. DLTs deﬁned as ≥Gr 3 non-hematologic toxicity except nausea, vomiting, or diarrhea that could be controlled by appropriate medical intervention or prophylaxis and that resolved within 48 hours, except electrolyte toxicities that can be corrected within 48 hours. Gr 3 rash attributed to the combination was considered a DLT if it remained Gr 3 despite maximal medical management for > 72 hours. Hematologic toxicities qualifying as DLTs included febrile neutropenia; Gr 4 neutropenia for > 7 days or thrombocytopenia < 25,000/mm3 (Gr 4) if associated with a bleeding event that did not result in hemodynamic instability but required an elective platelet transfusion; or a life-threatening bleeding event that resulted in urgent intervention and admission to an intensive care unit. Delay in starting cycle 2 of ≥14 days due to toxicity related to one or more protocol drugs was also considered a DLT. The ﬁrst 28-day cycle was considered the DLT period.
Time Frame: 28 days from the start of treatment.
Population: Two DLTs (Gr 3 maculopapular rash and Gr 3 hypophosphatemia) occurred at dose level 1.
Measure: Number; unit: participants
Arm/Group | Dose Level 1 - Onalespib IV 150 mg/m2 | Dose Level -1 - Onalespib IV 120 mg/m2
Number analyzed (Participants) | 3 | 8
participants | 2 | 0

2. Primary Outcome: Recommended Phase II Dose
Description: The maximum tolerated dose (MTD) of Onalespib IV in combination with 150 mg Erlotinib PO daily is based on toxicities observed during the first cycle and is defined as the highest dose tested in which fewer than 33% of patients experience an attributable DLT to the study drug, when at least 6 patients are treated at that dose and are evaluable for toxicity. Dose escalations proceeded according to a standard 3+3 design.
Time Frame: 28 days from start of treatment.
Measure: Number; unit: mg/m2
Groups:
- Treatment (Erlotinib Hydrochloride, Onalespib Lactate): Patients receive 150 erlotinib hydrochloride PO daily and starting dose of 150 mg/m2 onalespib lactate IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.
  Erlotinib Hydrochloride: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Onalespib Lactate: Given IV
  Pharmacological Study: Correlative studies
Arm/Group | Treatment (Erlotinib Hydrochloride, Onalespib Lactate)
Number analyzed (Participants) | 11
mg/m2 | 120

3. Primary Outcome: Number of Participants With Dose Limiting Toxicities.
Description: During the first course of therapy patients will be monitored for dose-limiting toxicities (DLT). Dose escalation will follow a 3+3 design, motivated by the desire to limit the incidence of dose-limiting toxicity to the lowest feasible levels and determine the recommended phase II dose. This outcome measure has been addressed in primary outcome measures 1 & 2.
Time Frame: Up to 4 weeks
Population: This outcome measure has been addressed in primary outcome measures 1 & 2.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level -1 - Onalespib IV 120 mg/m2: Patients receive 120 mg erlotinib hydrochloride PO daily and onalespib lactate IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.
  Erlotinib Hydrochloride: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Onalespib Lactate: Given IV
  Pharmacological Study: Correlative studies
Arm/Group | Dose Level 1 - Onalespib IV 150 mg/m2 | Dose Level -1 - Onalespib IV 120 mg/m2
Number analyzed (Participants) | 3 | 8
Participants | 2 | 0

4. Secondary Outcome: Number of Subject With Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to at least 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - Onalespib IV 150 mg/m2 | Dose Level -1 - Onalespib IV 120 mg/m2
Number analyzed (Participants) | 3 | 8
Participants | 0 | 0

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival will be summarized as time from first protocol treatment until progression or death from any cause, using the product-limit Kaplan-Meier estimator. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From start of treatment to time of progression or death from any cause, whichever occurs first, assessed up to at least 1 year
Population: The majority of patients (10/11) had lung cancers harboring EGFR ex20ins and were heavily pretreated.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Dose Level 1 - Onalespib IV 150 mg/m2: Patients receive 150 erlotinib hydrochloride PO daily and 150 mg/m2 of onalespib lactate IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.
  Erlotinib Hydrochloride: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Onalespib Lactate: Given IV
  Pharmacological Study: Correlative studies
Arm/Group | Dose Level 1 - Onalespib IV 150 mg/m2 | Dose Level -1 - Onalespib IV 120 mg/m2
Number analyzed (Participants) | 3 | 8
Months | NA [0.9 to NA] — NA - The Median and upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 4.5 [1.4 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

6. Secondary Outcome: Number of Subject With Overall Response (Recommended Phase II Dose)
Description: as for outcome 4
Time Frame: Up to at least 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Erlotinib Hydrochloride, Onalespib Lactate): Patients receive 150 erlotinib hydrochloride PO daily and 120 mg/m2 of onalespib lactate IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.
  Erlotinib Hydrochloride: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Onalespib Lactate: Given IV
  Pharmacological Study: Correlative studies
Arm/Group | Treatment (Erlotinib Hydrochloride, Onalespib Lactate)
Number analyzed (Participants) | 8
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 2 years and 4 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Dose Level 1 - Onalespib IV 150 mg/m2 | Dose Level -1 - Onalespib IV 120 mg/m2
All-Cause Mortality (participants affected / at risk) | 2/3 | 8/8
Serious Adverse Events (participants affected / at risk) | 3/3 | 3/8
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - Onalespib IV 150 mg/m2 (N=3) | Dose Level -1 - Onalespib IV 120 mg/m2 (N=8)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Expression aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - Onalespib IV 150 mg/m2 (N=3) | Dose Level -1 - Onalespib IV 120 mg/m2 (N=8)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 8 (35)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (10)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 3 (9) | 8 (60)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (10)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Chills (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (2) | 6 (25)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time pr (Investigations) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (2) | 3 (11)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 2 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (9)
Creatinine increased (Investigations) | 0 (0) | 3 (18)
INR increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (4) | 5 (18)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Serum amylase increased (Investigations) | 0 (0) | 1 (2)
Weight loss (Investigations) | 1 (1) | 4 (13)
White blood cell decreased (Investigations) | 1 (1) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 4 (11)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 5 (20)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (6)
Hyponatremia (Metabolism and nutrition disorders) | 3 (6) | 5 (19)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hand shaking (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
left shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 0 (0) | 2 (5)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (5)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
thoracic area (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (11)
Exfoliating skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail cracking (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (17)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (5)
cold sore (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
port site skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 3 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT02535338/Prot_SAP_000.pdf